CLINICAL TRIAL: NCT04709692
Title: An Open Label Phase 2a Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of (+)-SJ000557733 (SJ733) With or Without Cobicistat in Adult Patients With Acute, Uncomplicated Malaria Over a 42 Day Period
Brief Title: Efficacy of SJ733 in Adults With Uncomplicated Plasmodium Falciparum or Vivax Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R. Kiplin Guy (Other)
Collaborators: Global Health Innovative Technology Fund (Other); Eisai Inc. (Industry); Asociacion Civil Selva Amazonica (Other)
Responsible Party: Sponsor-Investigator, R. Kiplin Guy, Professor and Dean, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 53333
Record Dates: First submitted 2020-12-15; First posted 2021-01-14 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Malaria, Falciparum; Malaria, Vivax
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax | interventions — SJ733

STUDY DESIGN:
Intervention Model Description: There are 6 treatment arms (three cohorts, each with P. falciparum and P.vivax arms).Cohort progression will be managed independently for each treatment arm. Interim analysis will determine whether the data for each arm meets the success criteria
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Arm 1 A (cohort 1) (Other): Combination of 600 mg SJ733 with 150 mg Cobicistat administered orally once every day for three consecutive days for patients with P.vivax
  Interventions: Drug: (+)-SJ000557733 (SJ733)
- Arm 1 B (cohort 1) (Other): Combination of 600 mg SJ733 with 150 mg Cobicistat administered orally once every day for three consecutive days for patients with P.falciparum
  Interventions: Drug: (+)-SJ000557733 (SJ733)
- Arm 2 A (cohort 2) (Other): 600 mg SJ733 administered orally once every day for three consecutive days for patients with P.vivax
  Interventions: Drug: (+)-SJ000557733 (SJ733)
- Arm 2 B (cohort 2) (Other): 600 mg SJ733 administered orally once every day for three consecutive days for patients with P.falciparum
  Interventions: Drug: (+)-SJ000557733 (SJ733)
- Arm 3 A (cohort 3) (Other): Combination of 300 mg SJ733 with 150 mg Cobicistat administered orally once every day for three consecutive days for patients with P.vivax
  Interventions: Drug: (+)-SJ000557733 (SJ733)
- Arm 3 B (cohort 3) (Other): Combination of 300 mg SJ733 with 150 mg Cobicistat administered orally once every day for three consecutive days for patients with P.falciparum
  Interventions: Drug: (+)-SJ000557733 (SJ733)

INTERVENTIONS:
Drug: (+)-SJ000557733 (SJ733) — Anti-Malarial
  Other Names: SJ733

SUMMARY:
This Phase 2a trial recruits adult patients with uncomplicated P. vivax or P. falciparum blood-stage malaria mono-infection. The study drug SJ733 will be administered to examine its antimalarial efficacy, safety, and tolerability. This study also evaluates whether or not a fixed dose of the pharmacoenhancer cobicistat when given in combination with SJ733 significantly improves drug efficacy.

DETAILED DESCRIPTION:
This is an adaptive open label Phase 2a study to examine the antimalarial efficacy, safety, and tolerability of SJ733 in adult patients with uncomplicated P. vivax or P. falciparum blood-stage malaria monoinfection. SJ733 will be administered orally once every day for three consecutive days, with or without a fixed dose of the pharmacoenhancer cobicistat. The Phase 1 clinical data (completed under a US IND) and PK/PD models suggest that SJ733 is most likely to be curative as a 3-daily-dose pharmacoenhanced therapy, due to its moderately rapid clearance. There will be 1-3 cohorts with each cohort containing two treatment arms, P. falciparum (a) and P. vivax (b). Cohort progression will be managed independently for each treatment arm. Interim analysis will determine whether the data for a given treatment arm meets the success criteria, is inconclusive, or meets the failure criteria. Antimalarial efficacy will be examined over the period of 42 days. Additional aims are to characterize the safety and pharmacokinetics of SJ733. The results of this trial will identify active, well-tolerated doses for investigation in a larger Phase 2b clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 70 years of age (inclusive) at screening.
2. Body weight between 45 kg and 90 kg inclusive
3. Presence of mono-infection of P. falciparum or P. vivax confirmed by:

   1. Fever, as defined by axillary temperature ≥ 37.5°C or oral/rectal/tympanic temperature ≥ 38°C, or history of fever in the previous 24 hours (history of fever must be documented) and,
   2. Microscopically confirmed parasite infection: 1,000 to 40,000 asexual parasite count/µL blood
4. Written informed consent provided by participant, in accordance with local practice. If the participant is unable to write, witnessed consent is permitted according to local ethical considerations.
5. Ability to swallow oral medication.
6. Ability and willingness to participate and to comply with the study requirements
7. Agreement to hospitalization for at least 102 hours and/or until malarial parasites are not detected by microscopy on 2 consecutive occasions.
8. Agreement to come back to the hospital on Days 7, 10 or 11, 14, 17 or 18, 21, 24 or 25, 28, 35, and 42.
9. Women of child-bearing potential, has a negative pregnancy test at screening, and agrees to comply with one of the following during the treatment stage of the study and for a period of 90 days after stopping study drug:

   1. Use of oral, implantable, or injectable hormonal contraceptive, either combined or progestogen alone used in conjunction with barrier method as defined below.
   2. Use of an intrauterine device with a documented failure rate of <1% per year.
   3. Barrier method consisting of either condom or diaphragm.
   4. Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female.
   5. Complete abstinence from intercourse for 2 weeks prior to administration of study drug, throughout the study and for a period of 90 days after stopping study drug.

Exclusion Criteria:

1. Signs and symptoms of severe/complicated malaria according to the World Health Organization Criteria 2010 (Attachment 1: Definition of Severe Malaria)
2. Mixed Plasmodium infection.
3. Severe vomiting, defined as more than three times in the 24 hours prior to inclusion in the study, or severe diarrhea defined as 3 or more watery stools per day.
4. Severe malnutrition (defined as the weight-for-height being below -3 standard deviation or less than 70% of median of the NCHS/WHO normalized reference values)
5. Presence of a significant medical or psychiatric condition, or any other serious or chronic clinical condition requiring hospitalization, or any other condition that in the opinion of the investigator precludes participation in the study.
6. Female patients must not be either lactating or pregnant as demonstrated by a negative serum point-of-care pregnancy test pre-dose (the result of the pre-dose assessment must be confirmed negative prior to dosing).
7. Employment under the direct supervision of the investigators or study staff.
8. Clinically significant alterations to hematologic or clinical chemistry parameters that in the opinion of the investigator precludes participation in the study, including:

   1. AST/ALT > 3 x upper limit of normal range (ULN) and total bilirubin is normal
   2. AST/ALT > 2 x ULN and total bilirubin is >1 and <1.5 x ULN and conjugated bilirubin is > 35% of the total bilirubin
   3. Total bilirubin > 1.5 x ULN
   4. Serum creatinine levels > 2 x ULN
   5. Hb level < 8 g/dL
   6. Platelet level < 50,000/mm3
9. Participation in a clinical study of another investigational small molecule within 30 days or investigational biologic within 90 days prior to study enrollment or planning to begin such participation during the study.
10. Have received any antimalarial treatment (alone or in combination) in the past containing:

    1. Piperaquine, mefloquine, naphthoquine or sulphadoxine / pyrimethamine within the previous 6 weeks
    2. Amodiaquine or chloroquine within the previous 4 weeks
    3. Any artemisinin (artesunate, artemether, arteether or dihydroartemisinin) quinine, halofantrine, lumefantrine and any other anti-malarial treatment or antibiotics with antimalarial activity (including cotrimoxazole, tetracyclines, quinolones and fluoroquinolones, and azithromycin) within the past 14 days
11. Any medication from the list of prohibited medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro L Cuentas, MD, PhD, Principal Investigator — Asociación Civil Selva Amazónica (ACSA)
Locations (1):
- Asociación Civil Selva Amazónica (ACSA), Iquitos, Loreto, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jimenez-Diaz MB, Ebert D, Salinas Y, Pradhan A, Lehane AM, Myrand-Lapierre ME, O'Loughlin KG, Shackleford DM, Justino de Almeida M, Carrillo AK, Clark JA, Dennis AS, Diep J, Deng X, Duffy S, Endsley AN, Fedewa G, Guiguemde WA, Gomez MG, Holbrook G, Horst J, Kim CC, Liu J, Lee MC, Matheny A, Martinez MS, Miller G, Rodriguez-Alejandre A, Sanz L, Sigal M, Spillman NJ, Stein PD, Wang Z, Zhu F, Waterson D, Knapp S, Shelat A, Avery VM, Fidock DA, Gamo FJ, Charman SA, Mirsalis JC, Ma H, Ferrer S, Kirk K, Angulo-Barturen I, Kyle DE, DeRisi JL, Floyd DM, Guy RK. (+)-SJ733, a clinical candidate for malaria that acts through ATP4 to induce rapid host-mediated clearance of Plasmodium. Proc Natl Acad Sci U S A. 2014 Dec 16;111(50):E5455-62. doi: 10.1073/pnas.1414221111. Epub 2014 Dec 1. PMID 25453091
- [Background] Gaur AH, McCarthy JS, Panetta JC, Dallas RH, Woodford J, Tang L, Smith AM, Stewart TB, Branum KC, Freeman BB 3rd, Patel ND, John E, Chalon S, Ost S, Heine RN, Richardson JL, Christensen R, Flynn PM, Van Gessel Y, Mitasev B, Mohrle JJ, Gusovsky F, Bebrevska L, Guy RK. Safety, tolerability, pharmacokinetics, and antimalarial efficacy of a novel Plasmodium falciparum ATP4 inhibitor SJ733: a first-in-human and induced blood-stage malaria phase 1a/b trial. Lancet Infect Dis. 2020 Aug;20(8):964-975. doi: 10.1016/S1473-3099(19)30611-5. Epub 2020 Apr 8. PMID 32275867

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 B (Cohort 1): Combination of 600 mg SJ733 with 150 mg Cobicistat administered orally once every day for three consecutive days for patients with P.vivax
  (+)-SJ000557733 (SJ733): Anti-Malarial
- Arm 2 B (Cohort 2): 600 mg SJ733 administered orally once every day for three consecutive days for patients with P.vivax
  (+)-SJ000557733 (SJ733): Anti-Malarial
Period: Overall Study
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Started | 10 | 12
Completed | 10 | 11
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2) | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (12.47) | 42.9 (12.87) | 40.6 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 9 | 11 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  Peru | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Crude Adequate Clinical and Parasitological Response (ACPR)
Description: Crude Adequate Clinical and Parasitological Response (ACPR) defined as the absence of microscopically determined parasitemia (thick smear).
Time Frame: 14 days for each arm
Population: Only participants eligible for efficacy analysis were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 9
percentage of participants | 90 | 100

2. Primary Outcome: Percent of Patients With Treatment Related Adverse Events
Description: Number of and seriousness of treatment related adverse events as defined in Adult Toxicity Tables
Time Frame: 42 days for each arm
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 0 | 0

3. Primary Outcome: Percent of Patients With Clinically Significant Abnormal Laboratory Values
Description: Number of and seriousness of clinically significant abnormal laboratory values including changes from baseline in (biochemistry and hematology)
Time Frame: 42 days for each arm
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 0 | 2

4. Primary Outcome: Percent of Patients With Clinically Significant Abnormal Vital Signs
Description: Number of and seriousness of clinically significant abnormal vital signs including changes from baseline
Time Frame: 42 days for each arm
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 0 | 0

5. Primary Outcome: Percent of Patients With a Decrease in Hemoglobin (HB) > 2 g/dL From Baseline to an Absolute Value of < 5 g/dL
Description: Percent of patients with a decrease in hemoglobin (HB) > 2 g/dL from baseline to an absolute value of < 5 g/dL
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 0 | 0

6. Primary Outcome: Percent of Patients With an Absolute Neutrophil Count < 1,000/μL After Baseline
Description: Percent of patients with an absolute Neutrophil count < 1,000/μL after baseline
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 1 | 0

7. Primary Outcome: Percent of Patients Meeting Hy's Law Criteria
Description: Percent of patients meeting Hy's law criteria. Hy's law criteria: (1) Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevation of >3× the upper limit of normal (ULN); (2) total bilirubin (TBL) elevation of >2× ULN; (3) absence of initial findings of cholestasis (ie, absence of elevation of alkaline phosphatase [ALP] to >2× ULN); and (4) no other reason can be found to explain the combination of increased ALT and TBL, such as viral hepatitis A through E; other preexisting or acute liver disease; or another drug capable of causing the observed injury.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 0 | 0

8. Primary Outcome: Percent of Patients With Any ALT or AST ≥ 5 x ULN
Description: Percent of patients with Any ALT or AST ≥ 5 x upper limit of normal (ULN)
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 0 | 0

9. Primary Outcome: Percent of Patients With a ny AST or ALT ≥ 3 x ULN Together With the Appearance of Fatigue, Nausea, Vomiting, Right Upper Quadrant Pain or Tenderness, Fever, Rash and/or Eosinophilia
Description: Percent of patients with any AST or ALT ≥ 3 x ULN together with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (eosinophil percent or count above the upper limit of normal (ULN))
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 0 | 0

10. Primary Outcome: Percent of Patients With Persistent ALT ≥ 3 x ULN for a Period of More Than 4 Weeks.
Description: Percent of patients with persistent ALT ≥ 3 x ULN for a period of more than 4 weeks.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 0 | 0

11. Primary Outcome: Percent of Patients With Clinical Signs of Possible Cutaneous Adverse Reactions
Description: Percent of patients with clinical signs of possible cutaneous adverse reactions such as dermatitis, rash, erythematous rash, macular rash, papular rash, maculo-papular rash, pruritic rash, pustular rash, vesicular rash
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 0 | 0

12. Primary Outcome: Percent of Patients With Clinically Significant Increases in Venous Methemoglobin Levels
Description: Percent of patients with clinically significant increases in venous methemoglobin levels
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 0 | 0

13. Primary Outcome: Percent of Patients With Significant Changes in ECG Findings
Description: Percent of patients with significant changes in ECG findings, including heart rate, ECG intervals (PR, QTcB, QTcF), conduction changes or abnormalities
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Signs and Symptoms of Uncomplicated Malaria
Description: Number of participants with symptoms (including fever) or physical examination signs related to uncomplicated P. vivax or P. falciparum malaria
Time Frame: 42 days for each arm
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
Participants | 10 | 12

15. Secondary Outcome: Parasite Clearance Time
Description: Time to parasite clearance as measured by microscopy
Time Frame: 42 days for each arm
Population: Participants eligible for efficacy measurements were analyzed.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 9
hours | 15.60 [10.45 to 20.75] | 45.78 [15.83 to 75.73]

16. Secondary Outcome: Parasite Reduction Rate
Description: The parasite reduction rate is calculated as the slope of the linear portion of the regression fit of natural log of average parasitemia (per microliter) versus time (in hours). Reported slope is representative of all analyzed participants in each arm. Slope is analyzed during time frame in which there is active reduction of parasitemia by treatment (0->96 h).
Time Frame: 0->96 h, depending upon the time required to reach lower limit of detection
Population: Participants eligible for efficacy analysis were analyzed
Measure: Mean (95% Confidence Interval); unit: Ln(parasites/uL)/hour
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 9
Ln(parasites/uL)/hour | -0.33 [-0.39 to -0.27] | -0.08 [-0.09 to -0.06]

17. Secondary Outcome: Asexual Parasite Clearance Time
Description: Time to clearance of asexual parasites as measured by microscopy including half life of clearance. Clearance time represents the time at which the mean parasitemia has reached the given threshold for the arm/cohort. For PC100, the value represents the time at which all patients have undetectable parasitemia.
Time Frame: 42 days for each arm
Population: Only participants who were eligible for efficacy analysis were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 9
hours | 15.60 (8.32) | 45.78 (48.33)

18. Secondary Outcome: Percent Change in Asexual Parasites From Baseline
Description: Percentage change of asexual parasites as determined by microscopy, relative to baseline at the specified times. The value represents the average parasitemia in the arm/cohort at the given time (per microliter) versus time (in hours) compared to the average parasitemia at T0. Reported reduction is representative of all analyzed participants in each arm.
Time Frame: 42 days
Population: Only data from participants who were eligible for efficacy analysis were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change in parasites
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 9
percentage change in parasites
  Percent change in asexual parasites from baseline (24h) | -100 (0) | -97 (4.9)
  Percent change in asexual parasites from baseline (48h) | -100 (0) | -99.5 (1.5)
  Percent change in asexual parasites from baseline (72h) | -100 (0) | -99.8 (0.4)

19. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC)
Description: AUC of SJ733 and its metabolite SJ506 will be reported
Time Frame: 11 days for each arm
Population: Arm 2B participant whose condition worsened to severe malaria was not included in analysis due to no data available.
Measure: Median (95% Confidence Interval); unit: ug*h/L
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 11
ug*h/L
  AUC SJ733 at 24 hours | 110325 [43668.7 to 152576] | 24688.1 [14619.3 to 53068.5]
  AUC SJ506 at 24 hours | 14123.7 [10503.9 to 22190.3] | 31793.6 [20351.4 to 53646.8]
  AUC SJ733 at 48 hours | 271632.1 [110789.6 to 453783.7] | 56991.9 [32603.6 to 123993]
  AUC SJ506 at 48 hours | 29341.8 [25847.4 to 49196.8] | 74646.5 [45931.0 to 135353]
  AUC SJ733 at 72 hours | 450506.3 [183096.6 to 803489.9] | 92110.9 [51343.5 to 199588]
  AUC SJ506 at 72 hours | 46477.5 [42653.0 to 83301.5] | 118717 [72347.5 to 222926]
  AUC SJ733 at 96 hours | 517702.6 [203441.3 to 899838.3] | 105105.4 [55298.7 to 224240]
  AUC SJ506 at 96 hours | 73619.8 [59668.9 to 136436] | 134468 [79329.6 to 258502]
  AUC SJ733 at infinity | 538769.3 [207509.5 to 927069.4] | 111850 [56459.1 to 234779]
  AUC SJ506 at infinity | 93372.4 [65738.8 to 176802] | 141447 [82004.8 to 273535]

20. Secondary Outcome: Maximum Plasma Drug Concentration (Cmax)
Description: Cmax of SJ733 and its metabolite SJ506 will be reported
Time Frame: 11 days for each arm
Population: Arm 2B participant whose condition worsened to severe malaria was not included in analysis due to no data available.
Measure: Median (95% Confidence Interval); unit: ng/mL
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 11
ng/mL
  Cmax SJ733 | 9207.6 [3697.3 to 17736] | 2730.3 [1257.8 to 5032.7]
  Cmax SJ506 | 1244 [898.6 to 2424] | 2918.2 [1907.0 to 4602.0]

21. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Time to reach maximum plasma concentration (Tmax) of SJ733 will be reported
Time Frame: 11 days for each arm
Population: Arm 2B participant whose condition worsened to severe malaria was not included in analysis as there was no data available.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 11
hours | 53.97 [52.02 to 55.31] | 49.03 [48.57 to 55.12]

22. Secondary Outcome: Drug Clearance
Description: Drug clearance of SJ733 and its metabolite SJ506 will be reported
Time Frame: 11 days for each arm
Population: Arm 2B participant whose condition progressed to severe malaria was not included in analysis as no PK data was collected.
Measure: Median (95% Confidence Interval); unit: L/h
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 11
L/h
  CL SJ733 | 4.51 [3.14 to 15.69] | 16.06 [7.69 to 31.83]
  CL SJ506 | 19.49 [10.19 to 27.74] | 12.95 [6.68 to 22.41]

23. Secondary Outcome: Crude Adequate Clinical and Parasitological Response (ACPR) at Days 28, 35, and 42
Description: Crude Adequate Clinical and Parasitological Response (ACPR) at Days 28, 35, and 42 as measured by microscopy.
Time Frame: 42 days for each arm
Population: One participant from Arm 2b voluntarily withdrew from the study before the 14 day primary ACPR measurement. That participant's data is not included.
  One participant from Arm 2b developed severe malaria within hours after the first dose of SJ733. The participant received local treatment of standard of care for severe malaria. That participant's data is not included.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 10
percentage of participants
  ACPR day 28 | 20 | 30
  ACPR day 35 | 20 | 20
  ACPR day 42 | 20 | 10

24. Secondary Outcome: Time to Recurrence of Malaria Infection
Description: Time to recurrence of either P. vivax or P. falciparum malaria as measured by signs and symptoms or malaria and microscopy
Time Frame: 42 days for each arm
Population: Includes participants who were eligible for efficacy analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 9
days | 25.0 (9.51) | 24.1 (8.95)

25. Secondary Outcome: Fever Clearance Time
Description: Time from baseline to the first of two consecutive post-dose auxiliary temperature measurements < 37.5 C obtained within an interval of 4 to 24 hours of each other
Time Frame: 42 days for each arm
Population: Analysis includes all eligible participants, including (in arm 2B) one participant who developed severe malaria.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 12
hours | 9.200 [5.373 to 13.03] | 6.667 [4.004 to 9.329]

26. Other Pre Specified Outcome: Crude Adequate Clinical and Parasitological Response (ACPR), PCR Adjusted, at Days 7, 14, 28, 35, and 42
Description: Crude Adequate Clinical and Parasitological Response (ACPR) as adjusted by quantitative PCR of parasite DNA at Days 7, 14, 28, 35, and 42
Time Frame: 42 days for each arm
Population: Does not include Arm 2B participant who withdrew before day 14 nor Arm 2B participant who developed severe malaria and was treated with local standard of care for severe malaria.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 10
percentage of participants
  ACPR 7 | 100 | 100
  ACPR 14 | 80 | 80
  ACPR 28 | 20 | 30
  ACPR 35 | 20 | 20
  ACPR 42 | 20 | 10

27. Other Pre Specified Outcome: Time to Recurrence of Malaria Infection, PCR Adjusted
Description: Time to recurrence of either P. vivax or P. falciparum malaria as measured by PCR
Time Frame: 42 days for each arm
Population: Only participants eligible for efficacy analysis were analyzed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
Number analyzed (Participants) | 10 | 9
days | 24.0 (10.1) | 22.8 (9.94)

ADVERSE EVENTS:
Time Frame: AE data was collected for the 42 days that a participant was enrolled.
Description: A standard physical examination was performed as per the study schedule and included: general appearance, head and eyes, ears, nose and throat, chest and lungs, cardiovascular, abdomen, neurological, lymphatic, and musculoskeletal. Vital signs, body temperature, and ECGs were taken per the study schedule. Participants were given contact information to self-report AEs between study visits.
  Signs and symptoms of malaria were not recorded as adverse events.
Arm/Group | Arm 1 B (Cohort 1) | Arm 2 B (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/12
Other Adverse Events (participants affected / at risk) | 2/10 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 B (Cohort 1) (N=10) | Arm 2 B (Cohort 2) (N=12)
Febrile syndrome of probable viral etiology (Infections and infestations) | 1 (1) | 0 (0) — MedDRA code: 10072803 SAE due to Hospitalization - prolonged
Severe Malaria Grade 4 (Infections and infestations) | 0 (0) | 1 (1) — MedDRA: 10069722 Severe Malaria Grade 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 B (Cohort 1) (N=10) | Arm 2 B (Cohort 2) (N=12)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) — MedDRA: 10016952 Severity: mild
Hepatosplenomegaly (General disorders) | 1 (1) | 0 (0) — MedDRA: 10019847 Severity: Mild
Bilateral nephromegaly (Renal and urinary disorders) | 1 (1) | 0 (0) — MedDRA: 10048469 Severity: Mild
Alkaline Phosphatase Increase (Hepatobiliary disorders) | 0 (0) | 1 (1) — MedDRA: 10001675 Severity: Mild
Acute pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — MedDRA:10001002 Severity: Moderate
Increased Glucose (Endocrine disorders) | 0 (0) | 1 (1) — MedDRA: 10018421 Severity: Mild
Herpetic gingivostomatitis (Infections and infestations) | 0 (0) | 1 (1) — MedDRA: 10019996 Severity: Moderate

LIMITATIONS AND CAVEATS:
No participants were recruited into the P. falciparum arm as no participants who tested positive for P. falciparum met monoinfection inclusion criteria due to a decrease in P. falciparum monoinfection in the region.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. All data or results arising out of the performance of this Study shall be considered Information as defined above and shall not be used for the commercial benefit of Institution, Investigator, or Research Staff.
2. Any and all data resulting from the Study will not be presented or published in any form or media by the Institution, Investigator or Research Staff without the prior written consent of Sponsor which consent maybe as directed within the protocol.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT04709692/Prot_SAP_ICF_001.pdf